CLINICAL TRIAL: NCT00429676
Title: A Randomized Prospective Pilot Study Of Haloperidol In Addition To Standard Sedation In Mechanically Ventilated Patients With Delirium
Brief Title: Pilot Study of Haloperidol to Treat Critical Illness Delirium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Denver Health Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-0362
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2009-11

CONDITIONS: Delirium; Critical Illness
Keywords: Randomized; Controlled; Trial; Delirium; Haloperidol
MeSH Terms: conditions — Delirium; Critical Illness | interventions — Haloperidol

INTERVENTIONS:
Drug: Haloperidol

SUMMARY:
The goal of this study is to determine whether haloperidol reduces the time on the breathing machine in critically ill patients with delirium.

DETAILED DESCRIPTION:
Delirium is a frequent end-organ complication of critical illness and is an independent predictor of mortality in mechanically ventilated patients. However, management of delirium is a major therapeutic challenge and it is unknown if current therapies are disease modifying or function only as symptom management. Haloperidol has been demonstrated to reduce delirium in retrospective studies.

This study is a pilot prospective randomized clinical trial in the Denver Health Medical ICU to determine if haloperidol in addition to an evidence-based standard-of-care sedation protocol for the management of delirium results in a shortened duration of intubation and improvements in post-extubation cognitive status. The haloperidol dose is administered using titration-protocol guided by nursing assessment of delirium using the confusion assessment method for the ICU (CAM-ICU). The primary outcome is ventilator-free days out of the first 28, and secondary outcomes include duration of delirium, length and cost of hospitalization, 28-day mortality, usage of other sedatives, serum markers of delirium (neuron-specific enolase and protein S-100B), and cognitive-function scores at the time of ICU discharge, hospital discharge, and six-month follow-up.

The goal of the 20-patient pilot is demonstrating safety of the haloperidol protocol, as evaluated by an independent data-safety monitoring board. Following approval of the DSMB, 122 more patients will be enrolled in the full RCT to achieve power for an 80% chance of detecting a 40% decrease in duration of intubation with P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated within 24 hours of arrival to the ICU
* Delirium as assessed by CAM-ICU within 24 hours of arrival to the ICU
* Age > 18

Exclusion Criteria:

* Known allergy to haloperidol or other neuroleptics
* Neurological injury or trauma
* < 24 hours after a major operation
* History of Axis I psychiatric disorder or significant dementia
* Baseline QTc of > 500 msec or a pacemaker which makes the QTc uninterpretable
* History of seizure disorder
* Morbid obesity (> 1kg/cm body weight)
* Hepatic failure (Child's Class C)
* Neuromuscular disease (C5 or higher spinal cord injury, ALS, Guillain-Barre Syndrome, and myasthenia gravis)
* Malignancy or other irreversible disease or condition for which 6 month mortality is estimated to be ≥ 50%
* Pregnancy (negative pregnancy test required for women of child-bearing potential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days out of the first 28

SECONDARY OUTCOMES:
Duration of delirium
Length of hospitalization
Cost of hospitalization
28-day mortality
Usage of other sedatives
Serum markers of delirium (neuron-specific enolase and protein S-100B)
Cognitive-function scores at the time of ICU discharge, hospital discharge, and six-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ivor S Douglas, MD, Principal Investigator — University of Colorado Department of Pulmonary and Critical Care Medicine
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Milbrandt EB, Kersten A, Kong L, Weissfeld LA, Clermont G, Fink MP, Angus DC. Haloperidol use is associated with lower hospital mortality in mechanically ventilated patients. Crit Care Med. 2005 Jan;33(1):226-9; discussion 263-5. doi: 10.1097/01.ccm.0000150743.16005.9a. PMID 15644675